CLINICAL TRIAL: NCT00230685
Title: Hammersmith Hospital Patients With Pulmonary Arteriovenous Malformations (PAVMs) and Hereditary Haemorrhagic Telangiectasia
Brief Title: Case Notes Review on Patients With Hereditary Haemorrhagic Telangiectasia
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: The Margaret Hayton HHT Fund (Unknown)
Responsible Party: Sponsor
Other Study IDs: IC/CLS2
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic
Keywords: Pulmonary arteriovenous malformations
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This observational study is for individuals with Hereditary haemorrhagic telangiectasia and pulmonary arteriovenous malformations that are reviewed at the Hammersmith Hospital, London.

DETAILED DESCRIPTION:
The Hammersmith Hospital provides a clinical service for patients with Hereditary haemorrhagic telangiectasia and pulmonary arteriovenous malformations that is unique in the United Kingdom. Measurements obtained as part of standard clinical practice that has evolved since 1985 allow us to assess whether particular groups of individuals that we see are more prone to recognised complications such as strokes, brain abscesses, pregnancy related complications or pulmonary hypertension. We hypothesise that certain clinical characteristics will predict the susceptibility of individuals to particular complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending Hammersmith Hospital

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to the hereditary haemorrhagic telangiectasia clinical service at Hammersmith Hospital, imperial College Healthcare NHS Trust
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2000-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Stroke | Prospective
  Ischaemic stroke attributable to PAVMs
Venous thromboemboli (VTE) | Prospective
  VTE of any origin

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, Principal Investigator — Imperial College London
Locations (1):
- Respiratory Medicine, Hammersmith Hospital, London, United Kingdom

REFERENCES:
- [Result] Easey AJ, Wallace GM, Hughes JM, Jackson JE, Taylor WJ, Shovlin CL. Should asymptomatic patients with hereditary haemorrhagic telangiectasia (HHT) be screened for cerebral vascular malformations? Data from 22,061 years of HHT patient life. J Neurol Neurosurg Psychiatry. 2003 Jun;74(6):743-8. doi: 10.1136/jnnp.74.6.743. PMID 12754343
- [Result] Shovlin CL, Jackson JE, Bamford KB, Jenkins IH, Benjamin AR, Ramadan H, Kulinskaya E. Primary determinants of ischaemic stroke/brain abscess risks are independent of severity of pulmonary arteriovenous malformations in hereditary haemorrhagic telangiectasia. Thorax. 2008 Mar;63(3):259-66. doi: 10.1136/thx.2007.087452. Epub 2007 Nov 2. PMID 17981912
- [Result] Shovlin CL, Sulaiman NL, Govani FS, Jackson JE, Begbie ME. Elevated factor VIII in hereditary haemorrhagic telangiectasia (HHT): association with venous thromboembolism. Thromb Haemost. 2007 Nov;98(5):1031-9. PMID 18000608
- [Result] Shovlin CL, Sodhi V, McCarthy A, Lasjaunias P, Jackson JE, Sheppard MN. Estimates of maternal risks of pregnancy for women with hereditary haemorrhagic telangiectasia (Osler-Weber-Rendu syndrome): suggested approach for obstetric services. BJOG. 2008 Aug;115(9):1108-15. doi: 10.1111/j.1471-0528.2008.01786.x. Epub 2008 May 30. PMID 18518871
- [Result] Roked F, Jackson JE, Fuld J, Basheer FT, Chilvers ER, Beattie S, Shovlin CL. Pulmonary thromboemboli modifying the natural history of pulmonary arteriovenous malformations. Am J Respir Crit Care Med. 2011 Mar 15;183(6):828-9. doi: 10.1164/ajrccm.183.6.828. No abstract available. PMID 21471070
- [Result] Livesey JA, Manning RA, Meek JH, Jackson JE, Kulinskaya E, Laffan MA, Shovlin CL. Low serum iron levels are associated with elevated plasma levels of coagulation factor VIII and pulmonary emboli/deep venous thromboses in replicate cohorts of patients with hereditary haemorrhagic telangiectasia. Thorax. 2012 Apr;67(4):328-33. doi: 10.1136/thoraxjnl-2011-201076. Epub 2011 Dec 14. PMID 22169361
- [Result] Shovlin CL, Chamali B, Santhirapala V, Livesey JA, Angus G, Manning R, Laffan MA, Meek J, Tighe HC, Jackson JE. Ischaemic strokes in patients with pulmonary arteriovenous malformations and hereditary hemorrhagic telangiectasia: associations with iron deficiency and platelets. PLoS One. 2014 Feb 19;9(2):e88812. doi: 10.1371/journal.pone.0088812. eCollection 2014. PMID 24586400
- [Result] Shovlin CL, Tighe HC, Davies RJ, Gibbs JS, Jackson JE. Embolisation of pulmonary arteriovenous malformations: no consistent effect on pulmonary artery pressure. Eur Respir J. 2008 Jul;32(1):162-9. doi: 10.1183/09031936.00126207. Epub 2008 Apr 2. PMID 18385173
- [Result] Santhirapala V, Williams LC, Tighe HC, Jackson JE, Shovlin CL. Arterial oxygen content is precisely maintained by graded erythrocytotic responses in settings of high/normal serum iron levels, and predicts exercise capacity: an observational study of hypoxaemic patients with pulmonary arteriovenous malformations. PLoS One. 2014 Mar 17;9(3):e90777. doi: 10.1371/journal.pone.0090777. eCollection 2014. PMID 24637882
- [Result] Rizvi A, Macedo P, Babawale L, Tighe HC, Hughes JMB, Jackson JE, Shovlin CL. Hemoglobin Is a Vital Determinant of Arterial Oxygen Content in Hypoxemic Patients with Pulmonary Arteriovenous Malformations. Ann Am Thorac Soc. 2017 Jun;14(6):903-911. doi: 10.1513/AnnalsATS.201611-872OC. PMID 28267932
- [Result] Boother EJ, Brownlow S, Tighe HC, Bamford KB, Jackson JE, Shovlin CL. Cerebral Abscess Associated With Odontogenic Bacteremias, Hypoxemia, and Iron Loading in Immunocompetent Patients With Right-to-Left Shunting Through Pulmonary Arteriovenous Malformations. Clin Infect Dis. 2017 Aug 15;65(4):595-603. doi: 10.1093/cid/cix373. PMID 28430880
- [Result] Shovlin CL, Buscarini E, Hughes JMB, Allison DJ, Jackson JE. Long-term outcomes of patients with pulmonary arteriovenous malformations considered for lung transplantation, compared with similarly hypoxaemic cohorts. BMJ Open Respir Res. 2017 Oct 13;4(1):e000198. doi: 10.1136/bmjresp-2017-000198. eCollection 2017. PMID 29071074
- [Result] Thielemans L, Layton DM, Shovlin CL. Low serum haptoglobin and blood films suggest intravascular hemolysis contributes to severe anemia in hereditary hemorrhagic telangiectasia. Haematologica. 2019 Apr;104(4):e127-e130. doi: 10.3324/haematol.2018.205682. Epub 2018 Oct 18. No abstract available. PMID 30337360
- [Result] Fatania G, Gilson C, Glover A, Alsafi A, Jackson JE, Patel MC, Shovlin CL. Uptake and radiological findings of screening cerebral magnetic resonance scans in patients with hereditary haemorrhagic telangiectasia. Intractable Rare Dis Res. 2018 Nov;7(4):236-244. doi: 10.5582/irdr.2018.01103. PMID 30560015
- [Result] Gawecki F, Strangeways T, Amin A, Perks J, McKernan H, Thurainatnam S, Rizvi A, Jackson JE, Santhirapala V, Myers J, Brown J, Howard LSGE, Tighe HC, Shovlin CL. Exercise capacity reflects airflow limitation rather than hypoxaemia in patients with pulmonary arteriovenous malformations. QJM. 2019 May 1;112(5):335-342. doi: 10.1093/qjmed/hcz023. PMID 30657990
- [Result] Gawecki F, Myers J, Shovlin CL. Veterans Specific Activity Questionnaire (VSAQ): a new and efficient method of assessing exercise capacity in patients with pulmonary arteriovenous malformations. BMJ Open Respir Res. 2019 Mar 1;6(1):e000351. doi: 10.1136/bmjresp-2018-000351. eCollection 2019. PMID 30956797
- [Result] Shovlin CL, Millar CM, Droege F, Kjeldsen A, Manfredi G, Suppressa P, Ugolini S, Coote N, Fialla AD, Geisthoff U, Lenato GM, Mager HJ, Pagella F, Post MC, Sabba C, Sure U, Torring PM, Dupuis-Girod S, Buscarini E; VASCERN-HHT. Safety of direct oral anticoagulants in patients with hereditary hemorrhagic telangiectasia. Orphanet J Rare Dis. 2019 Aug 28;14(1):210. doi: 10.1186/s13023-019-1179-1. PMID 31462308
- [Result] Shovlin CL, Simeoni I, Downes K, Frazer ZC, Megy K, Bernabeu-Herrero ME, Shurr A, Brimley J, Patel D, Kell L, Stephens J, Turbin IG, Aldred MA, Penkett CJ, Ouwehand WH, Jovine L, Turro E. Mutational and phenotypic characterization of hereditary hemorrhagic telangiectasia. Blood. 2020 Oct 22;136(17):1907-1918. doi: 10.1182/blood.2019004560. PMID 32573726
- [Result] Anderson E, Sharma L, Alsafi A, Shovlin CL. Pulmonary arteriovenous malformations may be the only clinical criterion present in genetically confirmed hereditary haemorrhagic telangiectasia. Thorax. 2022 Jun;77(6):628-630. doi: 10.1136/thoraxjnl-2021-218332. Epub 2022 Feb 14. PMID 35165143
- [Result] Joyce KE, Onabanjo E, Brownlow S, Nur F, Olupona K, Fakayode K, Sroya M, Thomas GA, Ferguson T, Redhead J, Millar CM, Cooper N, Layton DM, Boardman-Pretty F, Caulfield MJ; Genomics England Research Consortium; Shovlin CL. Whole genome sequences discriminate hereditary hemorrhagic telangiectasia phenotypes by non-HHT deleterious DNA variation. Blood Adv. 2022 Jul 12;6(13):3956-3969. doi: 10.1182/bloodadvances.2022007136. PMID 35316832
- [Result] Shovlin CL, Almaghlouth FI, Alsafi A, Coote N, Rennie C, Wallace GM, Govani FS, Research Consortium GE. Updates on diagnostic criteria for hereditary haemorrhagic telangiectasia in the light of whole genome sequencing of 'gene-negative' individuals recruited to the 100 000 Genomes Project. J Med Genet. 2024 Jan 19;61(2):182-185. doi: 10.1136/jmg-2023-109195. No abstract available. PMID 37586837
- [Result] Mukhtar G, Shovlin CL. Unsupervised machine learning algorithms identify expected haemorrhage relationships but define unexplained coagulation profiles mapping to thrombotic phenotypes in hereditary haemorrhagic telangiectasia. EJHaem. 2023 Jul 3;4(3):602-611. doi: 10.1002/jha2.746. eCollection 2023 Aug. PMID 37601877
- [Result] Sharma L, Almaghlouth F, Mckernan H, Springett J, Tighe HC, Shovlin CL. Iron deficiency responses and integrated compensations in patients according to hereditary hemorrhagic telangiectasia ACVRL1, ENG and SMAD4 genotypes. Haematologica. 2024 Mar 1;109(3):958-962. doi: 10.3324/haematol.2022.282038. No abstract available. PMID 37731378